CLINICAL TRIAL: NCT00721396
Title: A Phase 2b, Open Label, Randomized, Parallel-Group, Multi-Center Study to Evaluate the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine When Administered With or Without Routine Infant Vaccinations to Healthy Infants According to Different Immunization Schedules.
Brief Title: Safety, Tolerability and Immunogenicity of Meningococcal B Recombinant Vaccine Administered With or Without Routine Infant Vaccinations to Healthy Infants According to Different Immunization Schedules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P12
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Meningococcal Infections
Keywords: Meningococcal disease,; Neisseria meningitidis serogroup B,; Prevention,; Vaccination,; Infants
MeSH Terms: conditions — Meningococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- B+R246 (Experimental): Subjects in this group received rMenB+OMV NZ vaccine at 2, 4, and 6 months of age, administered concomitantly with routine infant vaccinations.
  Interventions: Biological: rMenB+OMV NZ; Biological: combined diphtheria,tetanus,pertussis+polio+Hepatitis B+Haemophilus influenzae B vaccine; Biological: Pneumococcal vaccine
- B246_R357 (Experimental): Subjects in this group received rMenB+OMV NZ vaccine at at 2, 4, and 6 months of age; routine infant vaccinations were administered at 3, 5 and 7 months of age.
  Interventions: Biological: rMenB+OMV NZ; Biological: combined diphtheria,tetanus,pertussis+polio+Hepatitis B+Haemophilus influenzae B vaccine; Biological: Pneumococcal vaccine
- B+R234 (Experimental): Subjects in this group received rMenB+OMV NZ vaccine at 2, 3, 4 months of age, administered concomitantly with routine infant vaccinations.
  Interventions: Biological: rMenB+OMV NZ; Biological: combined diphtheria,tetanus,pertussis+polio+Hepatitis B+Haemophilus influenzae B vaccine; Biological: Pneumococcal vaccine
- R234 (Active Comparator): Subjects in this group received routine infant vaccines administered at 2, 3 and 4 months of age.
  Interventions: Biological: combined diphtheria,tetanus,pertussis+polio+Hepatitis B+Haemophilus influenzae B vaccine; Biological: Pneumococcal vaccine

INTERVENTIONS:
Biological: rMenB+OMV NZ
  Arms: B+R234; B+R246; B246_R357
Biological: combined diphtheria,tetanus,pertussis+polio+Hepatitis B+Haemophilus influenzae B vaccine
  Other Names: Infanrix Hexa
Biological: Pneumococcal vaccine
  Other Names: Prevenar

SUMMARY:
Primary :1.To demonstrate a sufficient immune response of rMenB+OMV NZ, when given concomitantly with routine infant vaccines to healthy infants at 2, 4 and 6 and 2, 3 and 4 months of age, as measured by percentage of subjects with serum bactericidal activity (SBA) titer ≥1:5, at 1 month after the third vaccination Secondary :To demonstrate that immunogenicity of routine infant vaccines, when given concomitantly with rMenB+OMV NZ to healthy infants at 2, 3 and 4 months of age, was non-inferior to that of routine infant vaccines given without rMenB+OMV NZ. 2. To demonstrate that the immunogenicity of rMenB+OMV NZ when given concomitantly with routine infant vaccines was non-inferior to that of rMenB+OMV NZ given without routine infant vaccines at 2, 4 and 6 months of age. 3. To assess prevalence of meningococcal B antibodies over the study period by evaluation of SBA, at baseline and at 1 month after third vaccination, in subjects- received routine infant vaccine without rMenB+OMV NZ.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month old infants (55-89 days, inclusive), who were born after full term pregnancy with an estimated gestational age ≥ 37 weeks and a birth weight ≥ 2.5 kg;
* For whom a parent/legal guardian has given written informed consent after the nature of the study has been explained.

Exclusion Criteria:

* History of any meningococcal B or C vaccine administration;
* prior vaccination with routine infant vaccines (Diphtheria, Tetanus, Pertussis, Polio, Haemophilus influenzae type b (Hib), and Pneumococcal antigens);
* Previous ascertained or suspected disease caused by N. meningitidis;
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component;
* Significant acute or chronic infection within the previous 7 days or axillary temperature major or equal to38 degrees within the previous day;
* Antibiotics within 6 days prior to enrollment;
* Any serious chronic or progressive disease;
* Known or suspected impairment or alteration of the immune system;
* Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation.

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1885 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (60):
- Belgium (6):
  - Novartis Investigational Site Nr. 59, Edegem, Antwerpen
  - Novartis Investigational Site Nr. 55, Antwerp, Antwerp
  - Study Investigational Site Nr. 60, Brussels, Brussels Capital
  - Novartis Investigational Site Nr. 57, Brussels, Brussels Capital
  - Novartis Investigational Site Nr. 56, Hasselt, Limburg
  - Novartis Investigational Site Nr. 58, Namur, Namur
- Czechia (4):
  - Novartis Investigational Site Nr. 95, Červený Kostelec, Hradec Králové
  - Novartis Investigational Site Nr. 93, Hradec Králové, Hradec Králové
  - Novartis Investigational Site Nr. 94, Pardubice, Pardubice
  - Novartis Investigational Site Nr. 96, Jindřichův Hradec, South Bohemian
- Germany (25):
  - Novartis Investigational Site Nr. 68, Bad Saulgau, Baden-Wurttemberg
  - Novartis Investigational Site Nr. 65, Bretten, Baden-Wurttemberg
  - Novartis Investigational Site Nr. 62, Kehl, Baden-Wurttemberg
  - Novartis Investigational Site Nr. 64, Oberstenfeld, Baden-Wurttemberg
  - Novartis Investigational Site Nr. 66, Welzheim, Baden-Wurttemberg
  - Novartis Investigational Site Nr. 69, Aschaffenburg, Bavaria
  - Novartis Investigational Site Nr. 71, Bremerhaven, City state Bremen
  - Novartis Investigational Site Nr. 72, Hamburg, Hamburg
  - Novartis Investigational Site Nr. 73, Baunatal, Hesse
  - Novartis Investigational Site Nr. 75, Bramsche, Lower Saxony
  - Novartis Investigational Site Nr. 85, Bielefeld, North Rhine-Westphalia
  - Novartis Investigational Site Nr. 81, Bochum, North Rhine-Westphalia
  - Novartis Investigational Site Nr. 79, Heiligenhaus, North Rhine-Westphalia
  - Novartis Investigational Site Nr. 80, Kleve Materborn, North Rhine-Westphalia
  - Novartis Investigational Site Nr. 78, Mönchengladbach, North Rhine-Westphalia
  - Novartis Investigational Site Nr. 82, Münster, North Rhine-Westphalia
  - Novartis Investigational Site Nr. 83, Warburg, North Rhine-Westphalia
  - Novartis Investigational Site Nr. 61, Mainz, Rhineland-Palatinate
  - Novartis Investigational Site Nr. 67, Schweigen, Rhineland-Palatinate
  - Novartis Investigational Site Nr. 86, Wanzleben, Saxony-Anhalt
  - Novartis Investigational Site Nr. 88, Itzenhoe, Schleswig-Holstein
  - Novartis Investigational Site Nr. 89, Itzenhoe, Schleswig-Holstein
  - Novartis Investigational Site Nr. 87, Stockelsdorf, Schleswig-Holstein
  - Novartis Investigational Site Nr. 70, Berlin, State of Berlin
  - Novartis Investigational Site Nr. 90, Erfurt, Thuringia
- Italy (5):
  - Novartis Investigational Site Nr. 5, Milan, Lombardy
  - Novartis Investigational Site Nr. 52, Milan, Lombardy
  - Novartis Investigational Site Nr. 6, Novara, Piedmont
  - Novartis Investigational Site Nr. 7, Florence, Tuscany
  - Novartis Investigational Site Nr. 9, Padua, Veneto
- Spain (16):
  - Novartis Investigational Site Nr. 46, Santiago de Compostela, A Coruña
  - Novartis Investigational Site Nr. 11, Almassora, Castellón
  - Novartis Investigational Site Nr. 10, Castellon, Castellón
  - Novartis Investigational Site Nr. 12, Vall D'Uixo, Castelló
  - Novartis Investigational Site Nr. 48, Vigo Pontevedra, Pontevedra
  - Novartis Investigational Site Nr. 49, Oviedo, Principality of Asturias
  - Novartis Investigational Site Nr. 25, Catarroja, Valencia
  - Novartis Investigational Site Nr. 21, L'Eliana, Valencia
  - Novartis Investigational Site 14, Sagunto, Valencia
  - Novartis Investigational Site Nr. 17, Valencia, Valencia
  - Novartis Investigational Site Nr. 24, Valencia, Valencia
  - Novartis Investigational Site Nr. 15, Valencia, Valencia
  - Novartis Investigational Site Nr. 18, Valencia, Valencia
  - Novartis Investigational Site Nr. 19, Valencia, Valencia
  - Novartis Investigational Site Nr. 16, Valencia, Valencia
  - Novartis Investigational Site Nr. 23, Valencia, Valencia
- United Kingdom (4):
  - Novartis Investigational Site Nr. 2, London, London
  - Novartis Investigational Site Nr. 1, Oxford, South East England
  - Novartis Investigational Site 3, Bristol, South West England
  - Novartis Investigational Site Nr. 4, Exeter, South West England

REFERENCES:
- [Derived] Zafack JG, Bureau A, Skowronski DM, De Serres G. Adverse events following immunisation with four-component meningococcal serogroup B vaccine (4CMenB): interaction with co-administration of routine infant vaccines and risk of recurrence in European randomised controlled trials. BMJ Open. 2019 May 19;9(5):e026953. doi: 10.1136/bmjopen-2018-026953. PMID 31110098
- [Derived] Gossger N, Snape MD, Yu LM, Finn A, Bona G, Esposito S, Principi N, Diez-Domingo J, Sokal E, Becker B, Kieninger D, Prymula R, Dull P, Ypma E, Toneatto D, Kimura A, Pollard AJ; European MenB Vaccine Study Group. Immunogenicity and tolerability of recombinant serogroup B meningococcal vaccine administered with or without routine infant vaccinations according to different immunization schedules: a randomized controlled trial. JAMA. 2012 Feb 8;307(6):573-82. doi: 10.1001/jama.2012.85. PMID 22318278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 centers in UK, 5 centers in Italy, 16 centers in Spain, 6 centers in Belgium, 25 centers in Germany and 4 centers in Czech Republic
Pre-assignment Details: All subjects enrolled were included in the trial.
Period: Overall Study
Arm/Group | B+R246 | B246_R357 | B+R234 | R234
Started | 627 | 628 | 318 | 312
Completed | 597 | 592 | 308 | 302
Not Completed | 30 | 36 | 10 | 10
Not completed — Adverse Event | 4 | 7 | 2 | 0
Not completed — Withdrawal by Subject | 12 | 15 | 3 | 7
Not completed — Lost to Follow-up | 7 | 9 | 3 | 3
Not completed — Protocol Violation | 4 | 3 | 1 | 0
Not completed — Inappropriate enrollment | 0 | 2 | 0 | 0
Not completed — Administrative reason | 3 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B+R246 | B246_R357 | B+R234 | R234 | Total
Number analyzed (Participants) | 627 | 628 | 318 | 312 | 1885
Age, Continuous [Mean (Standard Deviation); unit: days] | 68.7 (8.9) | 68.8 (9.4) | 68.8 (9.1) | 68.1 (9.0) | 68.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 292 | 312 | 164 | 159 | 927
  Male | 335 | 316 | 154 | 153 | 958

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Serum Bactericidal Activity ≥1:5 After Receiving Three Doses of rMenB+OMV NZ Vaccine
Description: The percentage of subjects with serum bactericidal activity(hSBA)titer ≥1:5 after receiving three doses of rMenB+OMV NZ vaccine were evaluated to demonstrate sufficient immune response following rMenB+OMV NZ vaccination, when given concomitantly with routine infant vaccines to healthy infants.
  The serum bactericidal antibodies directed against serogroup B meningococci, are measured by human complement Serum Bactericidal Assay (hSBA).
  The immune response was considered sufficient for groups B+R246 and B+R234 if the lower limit of the 2-sided 95% confidence interval was ≥ 70% for all three strains.
Time Frame: One month after third Men B vaccination
Population: The analysis was done on the Modified Intention to Treat (MIIT) population, ie, enrolled subjects who actually received a study vaccination and provided at least one evaluable serum sample after baseline.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B+R246 | B246_R357 | B+R234 | R234
Number analyzed (Participants) | 587 | 589 | 300 | 292
Percentages of subjects
  Baseline (44/76-SL strain)N=587,589,300,291 | 9 [6 to 11] | 7 [5 to 9] | 6 [4 to 10] | 6 [4 to 10]
  Post vaccination (44/76-SL)N=550,561,283,265 | 99 [98 to 100] | 99 [98 to 100] | 99 [97 to 100] | 4 [2 to 7]
  Baseline (5/99 strain)N=580,577,294,289 | 5 [4 to 8] | 7 [5 to 9] | 5 [3 to 8] | 6 [3 to 9]
  Post vaccination (5/99 strain)N=551,554,285,245 | 99 [98 to 100] | 99 [98 to 100] | 100 [99 to 100] | 5 [3 to 8]
  Baseline(NZ98/254 strain)N=582,583,298,292 | 3 [2 to 5] | 1 [0 to 2] | 2 [1 to 4] | 1 [0.083 to 2]
  Post vaccination(NZ98/254 strain)N=555,559,284,269 | 79 [75 to 82] | 87 [84 to 89] | 81 [76 to 85] | 4 [2 to 8]

2. Primary Outcome: Safety and Tolerability of 3 Doses of rMenB - Concomitantly With Routine Infant Vaccines at 2, 4 and 6 Months of Age - Concomitantly With Routine Vaccines at 2, 3 and 4 Months of Age - Alone at 2, 4 and 6 Months of Age
Description: Safety and Tolerability of 3 Doses of rMenB was assessed in terms of the number of subjects who reported solicited local and systemic adverse events when administered concomitantly with routine infant vaccines at 2,4,6 months of age (B+R246) to when rMenB+OMV NZ and routine vaccines were administered separately (group B246_R357).
Time Frame: 10 months (groups 1 and 2); 8 months (groups 3 and 4)
Population: All subjects receiving at least one injection and providing post-baseline safety data (Safety Set).
Measure: Number; unit: Number of subjects
Arm/Group | B+R246 | B246_R357 | B+R234 | R234
Number analyzed (Participants) | 624 | 627 | 318 | 311
Number of subjects
  Tenderness (N=624,626,318,311) | 529 | 491 | 265 | 0
  Erythema (N=624,626,318,311) | 506 | 516 | 257 | 0
  Induration (N=624,626,318,311) | 447 | 465 | 230 | 0
  Swelling (N=624,626,318,311) | 290 | 324 | 149 | 0
  Change in Eating Habits (N=624,626,318,311) | 470 | 473 | 249 | 159
  Sleepiness (N=624,626,318,311) | 523 | 525 | 282 | 224
  Vomiting (N=624,626,318,311) | 193 | 234 | 97 | 83
  Diarrhea (N=624,626,318,311) | 284 | 327 | 138 | 113
  Irritability (N=624,626,318,311) | 543 | 527 | 289 | 220
  Unusual Crying (N=624,626,318,311) | 526 | 515 | 268 | 186
  Rash (N=624,626,318,311) | 84 | 130 | 42 | 39
  Fever (≥38.0 C° %) ((N=624,627,318,311) | 501 | 447 | 243 | 160

3. Secondary Outcome: Non-inferiority of Immune Response to rMenB+OMV NZ Vaccination When Administered Concomitantly With Routine Infant Vaccines at 2,4,6 Months of Age
Description: The non-inferiority of immune response to rMenB+OMV NZ vaccination when administered concomitantly with routine infant vaccines at 2,4,6 months of age(B+R246) to when rMenB+OMV NZ and routine vaccines were administered separately (group B246_R357)was assessed in terms of percentage of subjects With hSBA≥ 1:5.
Time Frame: One month after 3rd Men B vaccination
Population: Analysis was done on the per-protocol population i.e all subjects in the MITT population who received all the relevant doses of vaccine correctly, provided evaluable serum samples at the relevant time points and had no major protocol violation as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B+R246 | B246_R357
Number analyzed (Participants) | 556 | 548
Percentages of subjects
  Baseline(44/76-SL strain) | 8 [6 to 11] | 7 [5 to 9]
  1 month post 3rd vaccination(44/76-SL)N=525,534 | 100 [99 to 100] | 100 [99 to 100]
  Baseline(5/99 strain)N=511,537 | 6 [4 to 8] | 7 [5 to 9]
  1 month post 3rd vaccination(5/99strain)N=527,529 | 100 [99 to 100] | 99 [98 to 100]
  Baseline(NZ98/254 strain)N=554,543 | 3 [2 to 5] | 1 [0 to 2]
  1 month post 3rd vaccination(NZ98/254 )N=530,534 | 79 [76 to 83] | 87 [84 to 90]
Statistical Analysis 1: Comparison: B+R246 vs B246_R357; Non-inferiority of immune responses against 44/76-SL strain when rMenB+OMV NZ vaccine was administered concomitantly with routine infant vaccines as compared to when rMenB+OMV NZ vaccine and routine vaccines were given separately; Test type: Non-Inferiority or Equivalence — Immune response of Group B+R246 was considered non-inferior to response of Group B246_R357, if at one month after the third rMenB+OMV NZ injection the 2-sided 95% lower confidence interval of the difference in the percentage of subjects with hSBA titer ≥1:5 was greater than -10% for each of the 3 strains; Miettinen and Nurminen method; Difference % (B+R246 minus B246_R357) = 0, 95% CI 2-sided [-1 to 1]
Statistical Analysis 2: Comparison: B+R246 vs B246_R357; Non-inferiority of immune responses against 5/99 strain when rMenB+OMV NZ vaccine was administered concomitantly with routine infant vaccines as compared to when rMenB+OMV NZ vaccine and routine vaccines were given separately; Test type: Non-Inferiority or Equivalence — Immune response of Group B+R246 was considered non-inferior to response of Group B246_R357, if at one month after the third rMenB+OMV NZ injection the 2-sided 95% lower confidence limit of the difference in the percentage of subjects with hSBA titer ≥5 was greater than -10% for each of the 3 strains; Miettinen and Nurminen method; Difference %(B+R246 minus B246_R357) = 0, 95% CI 2-sided [-1 to 1]
Statistical Analysis 3: Comparison: B+R246 vs B246_R357; Non-inferiority of immune responses against NZ98/254 strain when rMenB+OMV NZ vaccine was administered concomitantly with routine infant vaccines as compared to when rMenB+OMV NZ vaccine and routine vaccines were given separately; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 2]; Miettinen and Nurminen method; Difference % (B+R246 minus B246_R357) = -8, 95% CI 2-sided [-12 to -4]

4. Secondary Outcome: Non-inferiority of Immune Response to Diphtheria and Tetanus Antigens When Routine Vaccines Are Administered Concomitantly With rMen+OMV NZ Vaccine
Description: Non-inferiority of immune response to routine vaccine antigens when routine vaccines were administered concomitantly with rMenB+OMV NZ vaccine [group B+R234] to when only routine vaccines were given [Group R234] were assessed in terms of percentage of subjects with antibody concentrations ≥0.1 IU/mL against Diphtheria and Tetanus antigens as measured by enzyme-linked immunosorbent assay.
Time Frame: One month after 3rd vaccination
Population: All subjects in the Full Analysis Set/MITT population who received all the relevant doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to analysis: Per Protocol (PP) Population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B+R234 | R234
Number analyzed (Participants) | 269 | 259
Percentages of subjects
  Baseline (Diphtheria) | 25 [20 to 30] | 21 [16 to 26]
  1 month after 3rd vaccination(Diphtheria)N=261,232 | 100 [99 to 100] | 100 [98 to 100]
  Baseline (Tetanus) | 81 [76 to 86] | 86 [81 to 90]
  1 month after 3rd vaccination (Tetanus)N=261,232 | 100 [99 to 100] | 100 [98 to 100]
Statistical Analysis 1: Comparison: B+R234 vs R234; Non-inferiority of immune responses against Diphtheria antigen when routine vaccine was administered concomitantly with rMenB+OMV NZ vaccine to when only routine vaccines were administered; Test type: Non-Inferiority or Equivalence — Immune response of Group B+R234 was considered non-inferior to response of Group R234, if at one month after the third injection the 2-sided 95% lower confidence limit for the difference in the percentage of subjects with antibody response greater than the pre-specified cut off of for diphtheria (≥0.1 IU/mL) was >-10%; Miettinen and Nurminen method; Difference %(B+R234 minus R234) = 0, 95% CI 2-sided [-1 to 2]
Statistical Analysis 2: Comparison: B+R234 vs R234; Non-inferiority of immune response to Tetanus antigens when routine vaccines are administered concomitantly with rMen+OMV NZ vaccine; Test type: Non-Inferiority or Equivalence — Immune response of Group B+R234 was considered non-inferior to response of Group R234, if at one month after the third injection the 2-sided 95% lower confidence limit for the difference in the percentage of subjects with antibody response greater than the pre-specified cut off of for tetanus toxoid (≥0.1 IU/mL) was >-10%; Miettinen and Nurminen; Difference %(B+R234 minus R234) = 0, 95% CI 2-sided [-1 to 2]

5. Secondary Outcome: Geometric Mean Titers Against Neisseria Meningitidis Serogroup B, When rMenB+OMV NZ Vaccine is Administered Concomitantly With Routine Infant Vaccines.
Description: The hSBA antibody titers when rMenB+OMV NZ vaccine is administered concomitantly with routine infant vaccines to when rMenB+OMV NZ vaccine and routine vaccines were given separately are reported in terms of vaccine-group-specific geometric mean titers.
Time Frame: One month after third Men B vaccination
Population: PP Population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+R246 | B246_R357 | B+R234 | R234
Number analyzed (Participants) | 556 | 548 | 285 | 277
Titers
  Baseline (44/76-SL strain) N=556,548,285,277 | 1.49 [1.4 to 1.59] | 1.36 [1.28 to 1.46] | 1.34 [1.23 to 1.46] | 1.28 [1.19 to 1.37]
  post vaccination (44/76-SL) N=525,534,273,253 | 86 [80 to 92] | 113 [105 to 121] | 82 [75 to 91] | 1.16 [1.09 to 1.24]
  Baseline (5/99 strain) N=551,537,280,275 | 1.3 [1.21 to 1.39] | 1.28 [1.2 to 1.37] | 1.19 [1.09 to 1.3] | 1.24 [1.15 to 1.33]
  post vaccination (5/99 strain)N=527,529,275,236 | 537 [494 to 584] | 699 [643 to 759] | 325 [292 to 362] | 1.25 [1.08 to 1.45]
  Baseline (NZ98/254 strain)N=554,543,283,278 | 1.13 [1.08 to 1.18] | 1.08 [1.04 to 1.13] | 1.06 [1 to 1.12] | 1.07 [1.03 to 1.1]
  post vaccination (NZ98/254 strain)N=30,534,274,257 | 12 [11 to 14] | 18 [16 to 20] | 11 [9.14 to 12] | 1.11 [1.04 to 1.19]

6. Secondary Outcome: Geometric Mean Ratio of hSBA Titers, When rMenB+OMV NZ Vaccine is Administered Concomitantly With Routine Infant Vaccines.
Description: The geometric mean ratio(GMR) of GMTs at 1 month after 3rd rMenB+OMV NZ vaccination to prevaccination GMTs, when rMenB+OMV NZ was administered concomitantly with routine infant vaccines to when rMenB+OMV NZ vaccine and routine vaccines were given separately.
Time Frame: one month after third Men B vaccination
Population: PP Population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | B+R246 | B246_R357 | B+R234 | R234
Number analyzed (Participants) | 504 | 507 | 262 | 238
Ratio
  44/76-SL strain (N=501,507,262,236) | 58 [52 to 64] | 83 [74 to 92] | 61 [53 to 70] | 0.91 [0.83 to 1]
  5/99 strain (N=497,494,257,217) | 430 [379 to 487] | 553 [489 to 625] | 271 [231 to 318] | 1.03 [0.86 to 1.22]
  NZ98/254 strain (N=504,503,258,238) | 11 [9.28 to 12] | 16 [14 to 19] | 10 [8.52 to 12] | 1.05 [0.97 to 1.14]

7. Secondary Outcome: Percentage of Subjects With hSBA ≥1:8 After Receiving Three Doses of rMenB+OMV NZ Vaccine.
Description: The percentage of subjects with hSBA titers ≥1:8, following rMenB+OMV NZ vaccination when given concomitantly with routine infant vaccines to when rMenB+OMV NZ and routine vaccines were given separately.
Time Frame: One month after third Men B vaccination
Population: PP Population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B+R246 | B246_R357 | B+R234 | R234
Number analyzed (Participants) | 556 | 548 | 285 | 278
Percentages of subjects
  Baseline (44/76-SL strain)N=556,548,285,277 | 4 [3 to 6] | 3 [2 to 5] | 4 [2 to 7] | 2 [1 to 5]
  Post vaccination (44/76-SL)N=525,534,273,253 | 99 [98 to 100] | 100 [99 to 100] | 99 [97 to 100] | 2 [0 to 4]
  Baseline (5/99 strain)N=551,537,280,275 | 4 [2 to 6] | 3 [2 to 5] | 2 [1 to 5] | 4 [2 to 7]
  Post vaccination (5/99 strain)N=527,529,275,236 | 100 [99 to 100] | 99 [98 to 100] | 100 [99 to 100] | 3 [1 to 7]
  Baseline(NZ98/254 strain)N=554,543,283,278 | 1 [1 to 3] | 1 [0 to 2] | 1 [0.086 to 3] | 0.1 [0.0091 to 2]
  Post vaccination(NZ98/254 strain)N=530,534,274,257 | 67 [63 to 71] | 79 [75 to 82] | 69 [63 to 74] | 2 [1 to 5]

8. Secondary Outcome: Percentage of Subjects With 4-fold Rise in hSBA Titers, When rMenB+OMV NZ Vaccine is Administered Concomitantly With Routine Infant Vaccines.
Description: The percentage of subjects with 4-fold rise in hSBA titers at 1 month after 3rd rMenB+OMV NZ vaccination from baseline, when rMenB+OMV NZ was administered concomitantly with routine infant vaccines to when rMenB+OMV NZ vaccine and routine vaccines were given separately.
Time Frame: One month after third Men B vaccination
Population: PP Population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B+R246 | B246_R357 | B+R234 | R234
Number analyzed (Participants) | 504 | 507 | 262 | 238
Percentages of subjects
  44/76-SL strain (N=501,507,262,236) | 97 [96 to 99] | 99 [97 to 99] | 98 [96 to 99] | 1 [0 to 4]
  5/99 strain (N=497,494,257,217) | 99 [98 to 100] | 99 [98 to 100] | 100 [99 to 100] | 3 [1 to 7]
  NZ98/254 strain (N=504,503,258,238) | 66 [62 to 70] | 78 [74 to 81] | 69 [63 to 75] | 3 [1 to 5]

9. Secondary Outcome: Non-inferiority of Immune Response to Acellular Pertussis Antigens When Routine Vaccines Are Administered Concomitantly With rMen+OMV NZ Vaccine.
Description: Non-inferiority of immune response to routine vaccine antigens when routine vaccines were administered concomitantly with rMenB+OMV NZ vaccine [group B+R234] to when only routine vaccines were given [Group R234] were assessed in terms of percentage of subjects achieving seroconversion for pertussis antigens - Filamentous Hemagglutinin (FHA), Pertactin and Pertussis Toxoid (PT) at 1 month after 3rd vaccination versus baseline.
  Seroconversion was defined as a 4-fold increase for each pertussis antigen or in those initially seropositive, persistence of the pre-vaccination antibody concentration at least at the same antibody concentration as before vaccination, taking into account the decay of maternal antibodies.
Time Frame: 1 month after 3rd vaccination
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B+R234 | R234
Number analyzed (Participants) | 239 | 210
Percentages of subjects
  FHA | 94 [90 to 97] | 95 [91 to 97]
  Pertactin | 92 [88 to 95] | 95 [91 to 97]
  PT | 97 [94 to 99] | 98 [95 to 99]
Statistical Analysis 1: Comparison: B+R234 vs R234; Non-inferiority of immune responses against Pertussis antigen FHA when routine vaccine was administered concomitantly with rMenB+OMV NZ vaccine to when only routine vaccines were administered; Test type: Non-Inferiority or Equivalence — Group B+R234 was to be considered non-inferior to Group R234 if the 2-sided 95% lower confidence limit of this difference at 30 days after the last injection was greater than -10% for each of the antigens of the routine vaccinations; Miettinen and Nurminen method; Difference %(B+R234 minus R234) = -1, 95% CI 2-sided [-5 to 4]
Statistical Analysis 2: Comparison: B+R234 vs R234; Non-inferiority of immune responses against Pertussis antigen pertactin antigen when routine vaccine was administered concomitantly with rMenB+OMV NZ vaccine to when only routine vaccines were administered; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Difference %(B+R234 minus R234) = -2, 95% CI 2-sided [-7 to 2]
Statistical Analysis 3: Comparison: B+R234 vs R234; Non-inferiority of immune responses against Pertussis antigen PT when routine vaccine was administered concomitantly with rMenB+OMV NZ vaccine to when only routine vaccines were administered; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Difference %(B+R234 minus R234) = -1, 95% CI 2-sided [-4 to 2]

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs were collected for 7 days after each vaccination; SAEs, Medically attended AEs and AEs leading to premature withdrawal were collected throughout the study period.
Description: Of the 1885 enrolled subjects, 1882 received at least one vaccination and provided post-baseline safety data; these subjects were included in the safety analysis (B+R246 [625], B246_R357 [627], B+R234 [318], R234 [312]. Three subjects did not receive any vaccination and were excluded from the safety analysis (B+R246 [2], B246_R357 [1]).
Arm/Group | B+R246 | B246_R357 | B+R234 | R234
Serious Adverse Events (participants affected / at risk) | 63/625 | 57/627 | 19/318 | 19/312
Other Adverse Events (participants affected / at risk) | 620/625 | 623/627 | 316/318 | 305/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B+R246 (N=625) | B246_R357 (N=627) | B+R234 (N=318) | R234 (N=312)
Lymphadentitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Congenital musculoskeletal anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Craniosynostosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Urachal abnormality (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Retinal dystrophy (Eye disorders) | 0 | 0 | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Developmental delay (General disorders) | 1 | 1 | 0 | 0
Hyperpyrexia (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 4 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 2 | 3 | 2 | 3
Bronchitis (Infections and infestations) | 4 | 6 | 2 | 2
Bronchopneumonia (Infections and infestations) | 1 | 4 | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Enterovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Gatroenteritis (Infections and infestations) | 7 | 7 | 2 | 4
Gatroenteritis adenovirus (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0
Gatroenteritis rotavirus (Infections and infestations) | 1 | 1 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 0
Otitis media (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 3 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1 | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1 | 0
Staphylococcal bacteremia (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 1
Varicella (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 4 | 1 | 0 | 1
Accidental exposure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood alkaline phosphatase abnormal (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Crying (Nervous system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 2 | 0 | 1
Febrile convulsion (Nervous system disorders) | 1 | 2 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypotonic-hyporesponsive episode (Nervous system disorders) | 2 | 0 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 1 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Aponetic attack (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Prophylaxis (Surgical and medical procedures) | 0 | 1 | 0 | 0
Kawasaki's disease (Vascular disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B+R246 (N=625) | B246_R357 (N=627) | B+R234 (N=318) | R234 (N=312)
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 96 | 35 | 41
Somnolence (Nervous system disorders) | 523 | 525 | 282 | 224
Injection Site Induration (General disorders) | 489 | 519 | 254 | 204
Pyrexia (General disorders) | 514 | 462 | 246 | 176
Injection Site Erythema (General disorders) | 535 | 553 | 271 | 229
Injection Site Swelling (General disorders) | 328 | 383 | 170 | 115
Crying (General disorders) | 526 | 516 | 268 | 187
Injection Site Pain (General disorders) | 544 | 536 | 279 | 182
Irritability (Psychiatric disorders) | 543 | 527 | 289 | 220
Eating disorder (Psychiatric disorders) | 470 | 473 | 249 | 159
Diarrhea (Gastrointestinal disorders) | 302 | 338 | 145 | 123
Teething (Gastrointestinal disorders) | 30 | 51 | 7 | 13
Vomiting (Gastrointestinal disorders) | 208 | 245 | 100 | 85
Rash (Skin and subcutaneous tissue disorders) | 100 | 142 | 50 | 47
Eczema (Skin and subcutaneous tissue disorders) | 29 | 35 | 12 | 17
Nasopharyngitis (Infections and infestations) | 78 | 98 | 29 | 35
Rhinitis (Infections and infestations) | 67 | 91 | 28 | 36
Bronchitis (Infections and infestations) | 72 | 82 | 31 | 23
Upper Respiratory Tract Infection (Infections and infestations) | 76 | 72 | 24 | 16
Conjunctivitis (Infections and infestations) | 53 | 72 | 26 | 22
Viral Infection (Infections and infestations) | 42 | 53 | 17 | 26
Ear infection (Infections and infestations) | 48 | 52 | 15 | 14
Gastroenteritis (Infections and infestations) | 40 | 45 | 11 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days